CLINICAL TRIAL: NCT02850406
Title: A Phase 2a, Open-label, Single and Multiple Dose Study to Evaluate the Pharmacokinetics, Safety, Tolerability and Treatment Effect of GBT440 in Pediatric Participants With Sickle Cell Disease
Brief Title: Study to Evaluate the Effect of GBT440 in Pediatrics With Sickle Cell Disease
Acronym: HOPE-KIDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Emerging clinical data evaluated by Pfizer and shared with regulatory authorities indicates that the risk profile of voxelotor in people with SCD exceeds the benefits observed in previously generated global research and requires further assessment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GBT440-007; C5341020 (Other: Alias Study Number)
Expanded Access: NCT04724421 (No longer available)
Record Dates: First submitted 2016-07-01; First posted 2016-08-01 (Estimated); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Voxelotor (Experimental): Subjects to receive daily oral dosing of voxelotor according to which Part (A, B, C, or D), the subject is participating in:
  * Part A: Subjects to receive daily oral dosing of voxelotor for 1 day (single dose)
  * Part B: Subjects to receive daily oral dosing of voxelotor for up to 24 weeks (multiple dose)
  * Part C: Subjects to receive daily oral dosing of voxelotor for up to 48 weeks (1500mg or 1500mg equivalent dose)
  * Part D: Subjects to receive daily oral dosing of voxelotor for up to 48 weeks (1500mg equivalent dose)
  Interventions: Drug: Voxelotor

INTERVENTIONS:
Drug: Voxelotor — * Part A: Voxelotor will be administered as oral capsules or tablets
  * Part B: Voxelotor will be administered as oral capsules or tablets
  * Part C: Voxelotor will be administered as oral dispersible tablets or powder for oral suspension
  * Part D: Voxelotor will be administered as oral dispersible tablets or powder for oral suspension

SUMMARY:
This study consists of four parts, Parts A, B, C, and D.

* Part A is a single dose pharmacokinetic (PK) study in pediatric participants with Sickle Cell Disease ages 6 to 17 years.
* Part B is a multiple dose, safety, exploratory, efficacy, and PK study in adolescent participants with Sickle Cell Disease ages 12 to 17 years.
* Part C is a multiple dose, safety, tolerability, and PK study, which includes the assessment of hematological effects and the effect on TCD flow velocity of voxelotor in pediatric participants with Sickle Cell Disease ages 4 to 17 years.
* Part D is a multiple dose, safety, tolerability, and PK study, which examines the hematological effects of voxelotor in pediatric participants with Sickle Cell Disease ages 6 months to < 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with homozygous hemoglobin SS (HbSS) or hemoglobin S beta0 thalassemia (HbS β0thal)
* Age:

  * Part A - 6 to 17 years of age
  * Part B - 12 to 17 years of age
  * Part C - 4 to 17 years of age
  * Part D - 6 months to <4 years of age
* Hydroxyurea (HU) therapy:

  * Parts A, B, and C: A participant taking hydroxyurea (HU) may be enrolled if the dose has been stable for at least 3 months with no anticipated need for dose adjustment during the study and no sign of hematological toxicity.
  * Part D: A participant taking HU may be enrolled if the dose has been stable for at least 1 month. Titration to the maximum tolerated dose (MTD) is allowed during the study.
* Hemoglobin (HB):

  * Part A - No restriction
  * Parts B, C, & D - Hb ≤ 10.5 g/dL
* For Part C only: Participants 12 to 17 years of age must have a TCD velocity of ≥ 140 cm/sec measured anytime during screening.

Exclusion Criteria:

* Any one of the following requiring medical attention within 14 days of signing the Informed Consent Form (ICF):

  * Vaso-occlusive crisis (VOC)
  * Acute chest syndrome (ACS)
  * Splenic sequestration crisis
  * Dactylitis
* Requires chronic transfusion therapy
* History of stroke or meeting criteria for primary stroke prophylaxis (history of two TCD measurements ≥ 200 cm/sec by non-imaging TCD or ≥185 cm/sec by TCDi).
* Transfusion within 30 days prior to signing the ICF

Exclusion Criteria for Part D Only:

* Body weight <5 kg for 1 month prior to the screening visit and at the screening visit.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (13):
  - Brentwood Clinic UCSF Benioff Children's Hospital Oakland, Brentwood, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta Scottish Rite, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Illinois at Chicago Clinical Research Center, Chicago, Illinois
  - Our Lady of the Lake Children's Hospital (IP Address), Baton Rouge, Louisiana
  - Children's Mercy Hospital, Kansas City, Missouri
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - University Hospitals Cleveland Medical Center, Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- Lebanon (3):
  - American University of Beirut - Medical Center, Beirut
  - Rafik Hariri University Hospital, Beirut
  - Nini Hospital, Tripoli
- United Kingdom (4):
  - University College London Hospital, NHS Foundation Trust, London, Greater London
  - Barts Health NHS Trust, The Royal London Hospital, London
  - Guy's and St Thoma's NHS Foundation Trust, Evelina London Children's Hospital, London
  - Manchester University NHS Foundation Trust, Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Estepp JH, Kalpatthi R, Woods G, Trompeter S, Liem RI, Sims K, Inati A, Inusa BPD, Campbell A, Piccone C, Abboud MR, Smith-Whitley K, Dixon S, Tonda M, Washington C, Griffin NM, Brown C. Safety and efficacy of voxelotor in pediatric patients with sickle cell disease aged 4 to 11 years. Pediatr Blood Cancer. 2022 Aug;69(8):e29716. doi: 10.1002/pbc.29716. Epub 2022 Apr 21. PMID 35451176
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of four parts-Part A, B, C and D. The study was terminated as the emerging clinical data indicated that the risk profile of voxelotor in people with sickle cell disease (SCD) exceeded the benefits observed in previously generated global research and required further assessment.
Pre-assignment Details: A total of 147 pediatric participants with SCD (13 in Part A, 40 in Part B, 62 in Part C and 32 in Part D) were enrolled in the study.
Groups:
- Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg: Participants aged 12 to 17 years received a single oral dose of voxelotor 600 milligrams (mg) on Day 1.
- Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg: Participants aged 6 to 11 years received a single oral dose of voxelotor 600 mg on Day 1.
- Part B: Voxelotor 900 mg QD: Participants aged 12 to 17 years received once daily (QD) oral dose of voxelotor 900 mg for 24 weeks.
- Part B: Voxelotor 1500 mg QD: Participants aged 12 to 17 years received once daily oral dose of voxelotor 1500 mg for 24 weeks.
- Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD: Participants aged 4 to 11 years received once daily oral dose of voxelotor 1500 mg for 48 weeks.
- Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD: Participants aged 12 to 17 years received once daily oral dose of voxelotor 1500 mg for 48 weeks.
- Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD: Participants aged 6 months to <2 years received once daily oral dose of voxelotor 1500 mg for 48 weeks.
- Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD: Participants aged 2 to <4 years received once daily oral dose of voxelotor 1500 mg for 48 weeks.
Period: Part A (Up to 15 Days)
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Started | 7 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 7 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (Up to 28 Weeks)
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Started | 0 | 0 | 25 | 15 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 22 | 12 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Non compliance | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part C (Up to 52 Weeks)
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Started | 0 | 0 | 0 | 0 | 51 | 11 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 39 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 12 | 8 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 6 | 3 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Period: Part D (Up to 52 Weeks)
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 23
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population comprised of all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD | Total
Number analyzed (Participants) | 7 | 6 | 25 | 15 | 51 | 11 | 9 | 23 | 147
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.4 (0.79) | 8.2 (1.72) | 14.0 (1.68) | 13.9 (1.58) | 7.3 (2.06) | 13.1 (1.04) | 1.4 (0.41) | 3.0 (0.51) | 8.9 (4.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 11 | 10 | 27 | 4 | 3 | 9 | 71
  Male | 3 | 3 | 14 | 5 | 24 | 7 | 6 | 14 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 1 | 7
  Not Hispanic or Latino | 7 | 6 | 24 | 14 | 48 | 11 | 8 | 22 | 140
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Arab/Middle Eastern | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 3 | 3 | 18 | 11 | 44 | 11 | 5 | 9 | 104
  White | 2 | 2 | 6 | 4 | 3 | 0 | 2 | 9 | 28
  Multi-racial | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 5
  Middle Eastern or North African | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Part A: Maximum Concentration (Cmax) of Voxelotor in Whole Blood
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: Pharmacokinetic (PK) population comprised of all participants who received any amount of study drug and who provided PK data from at least one post-dose sample in plasma.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 7 | 6
Nanogram per milliliter | 24300 (36.39) | 47300 (43.62)

2. Primary Outcome: Part A: Area Under the Concentration-Time Curve (AUC) From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) of Voxelotor in Whole Blood
Description: AUC0-last was calculated using the linear/log trapezoid rule.
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: PK population comprised of all participants who received any amount of study drug and who provided PK data from at least one post-dose sample in plasma.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 7 | 6
Hours*nanogram per milliliter | 1570000 (38.13) | 2540000 (50.25)

3. Primary Outcome: Part A: Area Under the Concentration-Time Curve (AUC) From Time 0 Extrapolated to Infinity (AUC0-inf) of Voxelotor in Whole Blood
Description: AUC0-inf was calculated as AUCt + Ct/lambdaz, where AUCt=area under the concentration-time curve at designated time, Ct is the last quantifiable concentration for whole blood and lambdaz=elimination rate constant.
Time Frame: pre-dose, 2, 8, 24, 48, 96,168 and 336 hours post-dose
Population: PK population comprised of all participants who received any amount of study drug and who provided PK data from at least one post-dose sample in plasma. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 6 | 6
Hours*nanogram per milliliter | 1520000 (40.98) | 2570000 (50.59)

4. Primary Outcome: Part B: Change From Baseline to Week 24 in Hemoglobin Level
Time Frame: Baseline, Week 24
Population: Efficacy-Evaluable Population comprised of all participants who received any amount of study drug. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Gram per deciliter
Arm/Group | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD
Number analyzed (Participants) | 22 | 12
Gram per deciliter | 0.7 (0.86) | 0.2 (1.02)

5. Primary Outcome: Part C: Change From Baseline to Week 48 in Cerebral Blood Flow
Description: Cerebral blood flow was measured using transcranial Doppler (TCD) sonography. Change from baseline in cerebral blood flow as measured by the time-averaged mean of the maximum (TAMM) TCD velocity is reported.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Centimeter per second
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 34 | 3
Centimeter per second | -0.4 (16.76) | -26.3 (11.59)

6. Primary Outcome: Part D: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product during the course of a clinical investigation. TEAE was defined as an AE that emerged on or after initiation of study drug (having been absent pre-treatment), or an AE that existed pre-treatment and worsened on treatment (relative to the pre-treatment state) through 28 days after study drug discontinuation. An SAE was any AE that resulted in any of the following outcomes: death, life threatening adverse drug experience, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, congenital anomaly or birth defect, other important medical events. AEs were classified as SCD-related and non-SCD related.
Time Frame: From start of study treatment up to 28 days after study treatment discontinuation (Up to 52 weeks)
Population: Safety population comprised of all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 9 | 23
Participants
  Non-SCD related TEAEs | 9 | 20
  Non-SCD related SAEs | 6 | 12
  SCD related TEAEs | 6 | 14
  SCD related SAEs | 3 | 9

7. Secondary Outcome: Part A: Maximum Concentration (Cmax) of Voxelotor in Plasma
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 7 | 5
Nanogram per milliliter | 1880 (32.49) | 3390 (37.82)

8. Secondary Outcome: Part A: Maximum Concentration (Cmax) of Voxelotor in Red Blood Cells (RBC)
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 7 | 5
Nanogram per milliliter | 91500 (33.17) | 168000 (35.56)

9. Secondary Outcome: Part A: Area Under the Concentration-Time Curve (AUC) From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) of Voxelotor in Plasma
Description: AUC0-last was calculated using the linear/log trapezoid rule.
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 7 | 5
Hours*nanogram per milliliter | 104000 (20.85) | 148000 (38.69)

10. Secondary Outcome: Part A: Area Under the Concentration-Time Curve (AUC) From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) of Voxelotor in RBC
Description: AUC0-last was calculated using the linear/log trapezoid rule.
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 7 | 5
Hours*nanogram per milliliter | 6070000 (28.69) | 8950000 (47.05)

11. Secondary Outcome: Part A: Area Under the Concentration-Time Curve (AUC) From Time 0 Extrapolated to Infinity (AUC0-inf) of Voxelotor in Plasma
Description: AUC0-inf was calculated as AUCt + Ct/lambdaz, where AUCt=area under the concentration-time curve at designated time, Ct is the last quantifiable concentration for plasma and lambdaz is the elimination rate constant.
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 6 | 5
Hours*nanogram per milliliter | 101000 (20.51) | 150000 (38.01)

12. Secondary Outcome: Part A: Area Under the Concentration-Time Curve (AUC) From Time 0 Extrapolated to Infinity (AUC0-inf) of Voxelotor in RBC
Description: AUC0-inf was calculated as AUCt + Ct/lambdaz, where AUCt=area under the concentration-time curve at designated time, Ct is the last quantifiable concentration and lambdaz is the elimination rate constant.
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 4 | 5
Hours*nanogram per milliliter | 5550000 (24.31) | 9070000 (47.47)

13. Secondary Outcome: Part A: Time at Which Cmax Was Observed (Tmax) for Voxelotor in Whole Blood
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 7 | 6
Hours | 24.2 [7.67 to 49.9] | 8.73 [7.78 to 25.3]

14. Secondary Outcome: Part A: Time at Which Cmax Was Observed (Tmax) for Voxelotor in Plasma
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 7 | 5
Hours | 2.83 [1.95 to 9.00] | 2.83 [2.57 to 8.72]

15. Secondary Outcome: Part A: Time at Which Cmax Was Observed (Tmax) for Voxelotor in RBC
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 7 | 5
Hours | 9.00 [7.67 to 49.9] | 8.75 [8.72 to 25.3]

16. Secondary Outcome: Part A: Terminal Elimination Half-Life (T1/2) for Voxelotor in Whole Blood
Description: T1/2 was the time measured for the drug concentration to decrease by one half.
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 6 | 6
Hours | 31.9 (18.76) | 28.5 (26.18)

17. Secondary Outcome: Part A: Terminal Elimination Half-Life (T1/2) for Voxelotor in Plasma
Description: T1/2 was the time measured for the drug concentration to decrease by one half.
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 6 | 5
Hours | 46.4 (6.40) | 40.7 (31.48)

18. Secondary Outcome: Part A: Terminal Elimination Half-Life (T1/2) for Voxelotor in RBC
Description: T1/2 was the time measured for the drug concentration to decrease by one half.
Time Frame: pre-dose, 2, 8, 24, 48, 96, 168 and 336 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 4 | 5
Hours | 28.8 (12.89) | 27.3 (30.95)

19. Secondary Outcome: Part A: Percentage Hemoglobin (Hb) Occupancy
Description: Percentage hemoglobin occupancy (% Hb Occupancy) refers to the percentage of hemoglobin molecules within red blood cells that were bound to study drug. Concentration of voxelotor in whole blood and plasma was used to calculate %Hb occupancy. Percentage Hb occupancy within RBCs was estimated using the formula:
  ([Concentration of voxelotor in whole blood- {1-hematocrit}]*[Concentration of voxelotor in plasma/hematocrit])/5000*100.
Time Frame: 15 days
Population: Data was not collected as the model for Hb occupancy within RBCs was not developed for single dose administration (Part A). The model used to determine % Hb Occupancy was constructed via populational PK modelling and required data from multiple dose administration, thus cannot be applied to estimate the % Hb Occupancy for single doses.
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Part B: Percentage of Days With SCD Symptom Exacerbation During the First 24 Weeks of Treatment
Description: SCD symptoms were measured using the Patient Reported Outcome (PRO), Sickle Cell Disease Severity Measure (SCDSM) which was a self-administered 9-item questionnaire of SCD core symptoms including pain severity, frequency, and type, as well as fatigue and mental acuity, on a 4-point response scale that was completed daily using a handheld electronic device by the participants.
Time Frame: From Day 1 up to 24 weeks
Population: The variable represents a derivation from a new instrument developed by the sponsor specifically for this clinical program. Due to challenges in the validation of "Percentage of Days With SCD Symptom Exacerbation" from the instrument, specifically with the impact of missing data, the construct of this variable was not possible. A decision not to analyze this variable was documented in the statistical analysis plan.
Arm/Group | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Part B: Change From Baseline to Week 21 to 24 in the Sickle Cell Disease Severity Measure (SCDSM) Total Symptom Score (TSS)
Description: The SCDSM was a self-administered 9-item questionnaire of SCD core symptoms including pain severity, frequency, and type, as well as fatigue and mental acuity, on a 4-point response scale with a range of 0 (strongly disagree) to 4 (strongly agree) that was completed daily using a handheld electronic device by the participants. TSS was calculated as the sum of the 9-item questionnaire scores scaled to a 100-point scale with a range of 0 (no symptoms) to 100 (most severe symptoms). Baseline TSS was the average of the non-missing score during the Screening period. The average of change from baseline in SCDSM TSS score for the 4-week period (Week 21 to 24) is reported.
Time Frame: Baseline, Weeks 21 to 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD
Number analyzed (Participants) | 14 | 8
Units on a scale | 6.4 (17.98) | -10.7 (18.70)

22. Secondary Outcome: Part B: Percent Change From Baseline to Weeks 12 and 24 in Lactate Dehydrogenase (LDH)
Time Frame: Baseline, Weeks 12 and 24
Population: Efficacy-Evaluable Population comprised of all participants who received any amount of study drug. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD
Number analyzed (Participants) | 21 | 14
Percent change
  Week 12: number analyzed (Participants) | 19 | 14
  Week 12 | -6.3 (21.08) | -1.7 (32.78)
  Week 24: number analyzed (Participants) | 21 | 12
  Week 24 | -6.3 (22.47) | -1.9 (14.59)

23. Secondary Outcome: Part B: Percent Change From Baseline to Weeks 12 and 24 in Indirect Bilirubin
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD
Number analyzed (Participants) | 22 | 13
Percent change
  Week 12 | -32.1 (31.98) | -29.9 (33.59)
  Week 24: number analyzed (Participants) | 22 | 12
  Week 24 | -37.5 (29.07) | -32.1 (31.53)

24. Secondary Outcome: Part B: Percent Change From Baseline to Weeks 12 and 24 in Percentage Reticulocytes
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD
Number analyzed (Participants) | 23 | 14
Percent change
  Week 12 | -8.7 (36.46) | -3.5 (42.96)
  Week 24: number analyzed (Participants) | 22 | 12
  Week 24 | -14.1 (34.06) | 1.5 (43.18)

25. Secondary Outcome: Part B: Cmax of Voxelotor in Whole Blood and Plasma
Time Frame: Day 1 (pre-dose, 2, 8, 24 hours post-dose), pre-dose on Weeks 2, 4, 8, 12, 16, 20 and 24
Population: PK population comprised of participants who received at least one dose of voxelotor and had at least 1 measurable voxelotor concentration observation in plasma or whole blood with associated sampling time and dosing information.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD
Number analyzed (Participants) | 25 | 15
Microgram per milliliter
  Cmax, plasma | 5.64 (41) | 9.81 (37)
  Cmax, whole blood | 102 (38) | 159 (32)

26. Secondary Outcome: Part B: Area Under the Concentration-Time Curve (AUC) From Time 0 Extrapolated to Infinity (AUC0-inf) of Voxelotor for Whole Blood and Plasma
Description: as for outcome 12
Time Frame: Day 1 (pre-dose, 2, 8, 24 hours post-dose), pre-dose on Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD
Number analyzed (Participants) | 25 | 15
Hours*microgram per milliliter
  AUC0-inf, plasma | 113 (46) | 195 (40)
  AUC0-inf, whole blood | 2090 (43) | 3290 (36)

27. Secondary Outcome: Part B: Terminal Elimination Half-life of Voxelotor for Plasma and Whole Blood
Description: T1/2 was the time measured for the drug concentration to decrease by one half.
Time Frame: Day 1 (pre-dose, 2, 8, 24 hours post-dose), pre-dose on Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD
Number analyzed (Participants) | 25 | 15
Hours
  T1/2, plasma | 33 (41) | 33.9 (44)
  T1/2, whole blood | 31.1 (39) | 31.4 (41)

28. Secondary Outcome: Part B: Accumulation Ratio (Rac) of Voxelotor for Plasma and Whole Blood
Description: Accumulation ratio was calculated as ratio of area under the concentration-time curve from time 0 to 24 hours (AUC0-24) at steady-state (Day 28) to AUC0-24 on Day 1.
Time Frame: Day 1 (0 to 24 hours post-dose) and Day 28 (0 to 24 hours post-dose)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD
Number analyzed (Participants) | 25 | 15
Ratio
  Rac, plasma | 2.57 (29) | 2.62 (33)
  Rac, whole blood | 2.46 (27) | 2.47 (30)

29. Secondary Outcome: Part B: Percentage Hemoglobin Occupancy
Description: as for outcome 19
Time Frame: Day 28
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of bound hemoglobin
Arm/Group | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD
Number analyzed (Participants) | 25 | 15
Percentage of bound hemoglobin | 19.4 (34) | 29.5 (27)

30. Secondary Outcome: Part B: Change From Baseline to Week 12 and 24 in Cerebral Blood Flow
Description: Cerebral blood flow was measured using TCD sonography. Change from baseline in cerebral blood flow as measured by TAMM TCD velocity is reported.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Centimeter per second
Arm/Group | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD
Number analyzed (Participants) | 23 | 13
Centimeter per second
  Week 12 | 0.9 (16.48) | -0.1 (9.34)
  Week 24: number analyzed (Participants) | 20 | 12
  Week 24 | -2.1 (14.03) | 1.7 (14.26)

31. Secondary Outcome: Part C: Change From Baseline to Weeks 24 and 48 in Hemoglobin Level
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Grams per deciliter
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 41 | 6
Grams per deciliter
  Week 24 | 1.0 (1.16) | 0.8 (1.14)
  Week 48: number analyzed (Participants) | 37 | 3
  Week 48 | 0.7 (1.15) | -0.1 (0.20)

32. Secondary Outcome: Part C: Percent Change From Baseline to Weeks 24 and 48 in LDH
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 39 | 4
Percent change
  Week 24 | -5.1 (21.95) | -22.4 (22.08)
  Week 48: number analyzed (Participants) | 35 | 2
  Week 48 | -1.8 (23.80) | 3.9 (8.91)

33. Secondary Outcome: Part C: Percent Change From Baseline to Weeks 24 and 48 in Indirect Bilirubin
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 34 | 6
Percent change
  Week 24 | -36.9 (26.55) | -45.7 (24.93)
  Week 48: number analyzed (Participants) | 32 | 3
  Week 48 | -26.6 (37.05) | -33.0 (36.76)

34. Secondary Outcome: Part C: Percent Change From Baseline to Weeks 24 and 48 in Percentage Reticulocytes
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 37 | 5
Percent change
  Week 24 | -4.76 (42.999) | -1.17 (31.595)
  Week 48: number analyzed (Participants) | 34 | 2
  Week 48 | -0.33 (46.353) | 2.94 (38.295)

35. Secondary Outcome: Part C: Change From Baseline to Week 24 in Cerebral Blood Flow
Description: as for outcome 30
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Centimeter per second
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 40 | 6
Centimeter per second | -3.2 (15.69) | -11.8 (18.82)

36. Secondary Outcome: Part C: Time to Initial Hemoglobin Response
Description: Time to initial Hb response was defined as the time from first dose of study treatment to the first occurrence of a change from baseline in Hb > 1 gram per deciliter (g/dL).
Time Frame: From first dose of study treatment (Day 1) up to Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 36 | 8
Weeks | 4.9 (5.51) | 5.6 (4.90)

37. Secondary Outcome: Part C: Cmax of Voxelotor for Plasma and Whole Blood
Time Frame: Day 1 (15 minutes to 2 hours post-dose), pre-dose on Weeks 4, 8, 12, 16, 20, 24, 36 and 48
Population: PK population comprised of participants who received at least one dose of voxelotor and had at least 1 measurable voxelotor concentration observation in plasma or whole blood with associated sampling time and dosing information. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 49 | 11
Microgram per milliliter
  Cmax, plasma | 7.83 (61) | 9.04 (43)
  Cmax, whole blood | 127 (52) | 137 (38)

38. Secondary Outcome: Part C: Area Under the Concentration-Time Curve (AUC) From Time 0 Extrapolated to Infinity (AUC0-inf) of Voxelotor for Whole Blood and Plasma
Description: as for outcome 12
Time Frame: Day 1 (15 minutes to 2 hours post-dose), pre-dose on Weeks 4, 8, 12, 16, 20, 24, 36 and 48
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 49 | 11
Hours*microgram per milliliter
  AUC0-inf, plasma | 160 (72) | 184 (44)
  AUC0-inf, whole blood | 2660 (64) | 2880 (41)

39. Secondary Outcome: Part C: Terminal Elimination Half-life (T1/2) of Voxelotor for Whole Blood and Plasma
Description: T1/2 was the time measured for the drug concentration to decrease by one half.
Time Frame: Day 1 (15 minutes to 2 hours post-dose), pre-dose on Weeks 4, 8, 12, 16, 20, 24, 36 and 48
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 49 | 11
Hours
  T1/2, plasma | 41.6 (50) | 35.6 (28)
  T1/2, whole blood | 37.4 (48) | 32.7 (25)

40. Secondary Outcome: Part C: Percentage Hemoglobin Occupancy of Voxelotor
Description: as for outcome 19
Time Frame: Day 28
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of bound hemoglobin
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 49 | 11
Percentage of bound hemoglobin | 24.7 (47) | 27.7 (30)

41. Secondary Outcome: Part C: Percentage of Participants With Normal Transcranial Doppler (TCD) Flow Velocity at Week 48
Description: Normal TCD flow velocity was considered as < 170 centimeter per second (cm/sec) by non-imagining TCD or < 155 cm/sec by imaging transcranial Doppler (TCDi). Percentage of participants with normal TCD flow velocity at Week 48 by Baseline TCD group (i.e. Baseline normal TCD [<170 cm/sec] and Baseline conditional TCD [>=170 cm/sec] is reported.
Time Frame: Week 48
Population: Efficacy-Evaluable Population comprised of all participants who received any amount of study drug. All participants reported under, 'Overall Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for each row. Here, 'Number Analyzed ' signifies number of participants evaluable for each row.
Measure: Number; unit: Percentage of participants
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 34 | 3
Percentage of participants
  Baseline normal: number analyzed (Participants) | 27 | 1
  Baseline normal | 96.3 [lower limit 15.69] | 100 [lower limit 18.82]
  Baseline conditional: number analyzed (Participants) | 7 | 2
  Baseline conditional | 42.9 | 100

42. Secondary Outcome: Part C: Annualized Incidence Rate of Vaso-occlusive Crisis (VOC) Events
Description: VOC events included preferred terms of sickle cell anaemia with crisis, acute chest syndrome, pneumonia necrotising and pneumonia. Annualized incidence rate was calculated as total number of events divided by total person years. Total person years=sum of participants treatment period in years, which covered the time from first dose to last dose.
Time Frame: Up to Week 48
Population: Efficacy-Evaluable Population comprised of all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: VOC events per person year
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 51 | 11
VOC events per person year | 1.246 [0.912 to 1.662] | 2.250 [1.123 to 4.025]

43. Secondary Outcome: Part C: Annualized Incidence Rate of Stroke Events
Description: Annualized incidence rate was calculated as total number of events divided by total person years. Total person years=sum of participants treatment period in years, which covered the time from first dose to last dose.
Time Frame: Up to Week 48
Population: Efficacy-Evaluable Population comprised of all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Stroke events per person year
Arm/Group | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 51 | 11
Stroke events per person year | 0.000 [0.000 to 0.100] | 0.000 [0.000 to 0.754]

44. Secondary Outcome: Part D: Cmax of Voxelotor for Plasma and Whole Blood
Time Frame: Day 1 (anytime between 15 minutes to 2 hours post-dose), pre-dose on Weeks 2, 8, 12, 16, 24, 36 and 48
Population: PK population comprised of participants who received at least one dose of voxelotor and had at least 1 measurable voxelotor concentration observation in plasma or whole blood with associated sampling time and dosing information. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 8 | 21
Microgram per milliliter
  Cmax, plasma | 5.01 (73) | 9.45 (34)
  Cmax, whole blood | 87.2 (74) | 149 (30)

45. Secondary Outcome: Part D: Area Under the Concentration-Time Curve (AUC) From Time 0 Extrapolated to Infinity (AUC0-inf) of Voxelotor for Plasma and Whole Blood
Description: as for outcome 12
Time Frame: Day 1 (anytime between 15 minutes to 2 hours post-dose), pre-dose on Weeks 2, 8, 12, 16, 24, 36 and 48
Population: as for outcome 44
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 8 | 21
Hours*microgram per milliliter
  AUC0-inf, plasma | 89.9 (110) | 186 (38)
  AUC0-inf, whole blood | 1600 (120) | 3040 (36)

46. Secondary Outcome: Part D: T1/2 of Voxelotor for Plasma and Whole Blood
Description: T1/2 was the time measured for the drug concentration to decrease by one half.
Time Frame: Day 1 (anytime between 15 minutes to 2 hours post-dose), pre-dose on Weeks 2, 8, 12, 16, 24, 36 and 48
Population: as for outcome 44
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 8 | 21
Hours
  T1/2, plasma | 24.1 (70) | 36.1 (40)
  T1/2, whole blood | 21.7 (82) | 32.7 (38)

47. Secondary Outcome: Part D: Percentage Hemoglobin Occupancy
Description: as for outcome 19
Time Frame: Day 28
Population: as for outcome 44
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of bound hemoglobin
Arm/Group | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 8 | 21
Percentage of bound hemoglobin | 17.5 (60) | 28.9 (26)

48. Secondary Outcome: Part D: Change From Baseline to Weeks 24 and 48 in Hemoglobin Level
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Grams per deciliter
Arm/Group | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 7 | 20
Grams per deciliter
  Week 24 | 0.4 (2.03) | 0.6 (1.02)
  Week 48 | 0.5 (1.53) | 0.7 (1.45)

49. Secondary Outcome: Part D: Percent Change From Baseline to Weeks 24 and 48 in LDH
Time Frame: Baseline, Weeks 24 and 48
Population: Efficacy-Evaluable Population comprised of all participants who received any amount of study drug. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 6 | 20
Percent change
  Week 24 | 27.6 (56.46) | -0.4 (31.53)
  Week 48: number analyzed (Participants) | 6 | 18
  Week 48 | 26.3 (43.98) | 7.4 (45.94)

50. Secondary Outcome: Part D: Percent Change From Baseline to Weeks 24 and 48 in Indirect Bilirubin
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 7 | 18
Percent change
  Week 24 | -14.4 (28.11) | -24.5 (24.50)
  Week 48: number analyzed (Participants) | 7 | 17
  Week 48 | 4.4 (42.05) | -24.5 (21.97)

51. Secondary Outcome: Part D: Percent Change From Baseline to Weeks 24 and 48 in Reticulocytes Count
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 6 | 14
Percent change
  Week 24 | -3.6 (28.64) | 3.8 (31.88)
  Week 48: number analyzed (Participants) | 6 | 13
  Week 48 | -11.5 (31.19) | -0.7 (29.70)

52. Secondary Outcome: Part D: Time to Initial Hemoglobin Response
Description: Time to initial Hb response, defined as the time from first dose of study treatment to the first occurrence of a change from baseline in Hb > 1 g/dL.
Time Frame: From first dose of study treatment (Day 1) up to Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 6 | 18
Weeks | 8.0 (7.60) | 4.7 (8.80)

53. Secondary Outcome: Part D: Annualized Incidence Rate of VOC Events
Description: VOC events included preferred terms of 'Sickle cell anemia with crisis', 'Acute chest syndrome', 'Pneumonia necrotising,' and 'Pneumonia. Annualized incidence rate was calculated as total number of events divided by total person years. Total person years=sum of participants treatment period in years, which covered the time from first dose to last dose.
Time Frame: Up to Week 48
Population: Efficacy-Evaluable Population comprised of all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: VOC events per person year
Arm/Group | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 9 | 23
VOC events per person year | 1.473 [0.706 to 2.708] | 1.399 [0.914 to 2.050]

54. Secondary Outcome: Part D: Annualized Incidence Rate of Stroke Events
Description: as for outcome 43
Time Frame: Up to Week 48
Population: Efficacy-Evaluable Population comprised of all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Stroke events per person year
Arm/Group | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
Number analyzed (Participants) | 9 | 23
Stroke events per person year | 0.000 [0.000 to 0.543] | 0.000 [0.000 to 0.198]

ADVERSE EVENTS:
Time Frame: Part A: From start of treatment on Day 1 up to 2 weeks after last dose (up to Day 15); Part B, C and D: From start of treatment on Day 1 up to 4 weeks after last dose (up to Week 28 for Part B and up to Week 52 for Parts C and D).
Description: An AE term may be reported as both serious and non-serious AE but are distinct events. An AE may be serious for 1 participant and non-serious for another participant, or a participant may have experienced both a serious and non-serious episode of the same event. Safety population comprised of all participants who received any amount of study drug.
Arm/Group | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg | Part B: Voxelotor 900 mg QD | Part B: Voxelotor 1500 mg QD | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/25 | 0/15 | 0/51 | 0/11 | 0/9 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/6 | 12/25 | 7/15 | 23/51 | 8/11 | 7/9 | 14/23
Other Adverse Events (participants affected / at risk) | 6/7 | 3/6 | 22/25 | 15/15 | 46/51 | 11/11 | 9/9 | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg (N=7) | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg (N=6) | Part B: Voxelotor 900 mg QD (N=25) | Part B: Voxelotor 1500 mg QD (N=15) | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD (N=51) | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD (N=11) | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD (N=9) | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD (N=23)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 0 | 9 | 4 | 18 | 7 | 1 | 7 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Hemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Priapism (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 8 | 0 | 1 | 2 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 3 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 5 | 1 | 2 | 3 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Hypersplenism (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 3 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Platelet disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Periorbital swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Ultrasound head abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Splenectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Participants Aged 12 to 17 Years: Voxelotor 600 mg (N=7) | Part A: Participants Aged 6 to 11 Years: Voxelotor 600 mg (N=6) | Part B: Voxelotor 900 mg QD (N=25) | Part B: Voxelotor 1500 mg QD (N=15) | Part C: Participants Aged 4 to 11 Years: Voxelotor 1500 mg QD (N=51) | Part C: Participants Aged 12 to 17 Years: Voxelotor 1500 mg QD (N=11) | Part D: Participants Aged 6 Months to <2 Years: Voxelotor 1500 mg QD (N=9) | Part D: Participants Aged 2 to <4 Years: Voxelotor 1500 mg QD (N=23)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 1 | 5 | 3 | 10 | 2 | 5 | 10 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Priapism (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Nausea (Gastrointestinal disorders) | 2 | 0 | 9 | 3 | 4 | 1 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 4 | 3 | 5 | 1 | 1 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Vomiting (Gastrointestinal disorders) | 0 | 0 | 5 | 2 | 15 | 1 | 5 | 2 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 10 | 1 | 2 | 3 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 2 | 0 | 1 | 2 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 2 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 10 | 3 | 7 | 0 | 2 | 4 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 4 | 3 | 2 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 4 | 1 | 2 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Viral infection (Infections and infestations) | 0 | 0 | 5 | 0 | 7 | 0 | 2 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 2 | 8 | 2 | 2 | 7 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Body tinea (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Headache (Nervous system disorders) | 1 | 0 | 7 | 4 | 9 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Non-cardiac chest pain (General disorders) | 1 | 0 | 2 | 2 | 1 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Pyrexia (General disorders) | 0 | 0 | 2 | 2 | 15 | 2 | 4 | 8 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Pain (General disorders) | 0 | 0 | 2 | 1 | 4 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 3 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 2 | 2 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 6 | 0 | 1 | 2 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Reticulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Transaminases increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Bacterial test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Stress (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Retinopathy sickle cell (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Tinea faciei (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Tonsillar erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Influenza A virus test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Left atrial dilatation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Sports injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Epiphyseal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Albuminuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Allergic oedema (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Encopresis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Enuresis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Hypersplenism (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Viral rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Ultrasound head abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Foreign body ingestion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Benign lymph node neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms
Allergic respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v19.1 for Part A and Part B arms, MedDRA v25.1 for Part C arms and MedDRA v26.0 for Part D arms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT02850406/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT02850406/SAP_001.pdf